CLINICAL TRIAL: NCT03137017
Title: A Relative Bioavailability Trial to Investigate the Pharmacokinetics of Two Immediate Release Fixed Dose Combinations of Hydrocodone Bitartrate and Acetaminophen (a New Abuse Deterrent Tablet and a Marketed Tablet) Administered Under Fasted and Fed Conditions in Healthy Male and Female Adult Subjects
Brief Title: A Comparison of Plasma Concentrations of Hydrocodone and Acetaminophen After Administration of a New and a Marketed Tablet Formulation Under Fasted and Fed Conditions in Healthy Adults
Status: Withdrawn | Phase: Phase 1 | Type: Interventional
Why Stopped: program discontinued
Sponsor: Grünenthal GmbH (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: HP7014-01; U1111-1183-5343 (Other: World Health Organization)
Record Dates: First submitted 2017-04-27; First posted 2017-05-02 (Actual); Last update posted 2017-07-21 (Actual); Status verified 2017-07

CONDITIONS: Opioid-Related Disorders; Pain, Acute; Pain, Postoperative
Keywords: Abuse deterrent formulation; Hydrocodone; Analgesics, Opioid; Narcotics
MeSH Terms: conditions — Opioid-Related Disorders; Acute Pain; Pain, Postoperative | interventions — oxycodone-acetaminophen; Hydrocodone; Acetaminophen

STUDY DESIGN:
Intervention Model Description: The randomization will be realized using a Williams Square with a 4x4 design.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (4):
- GRT7014 fasted (Experimental): Abuse deterrent formulation of a fixed dose combination of hydrocodone bitartrate 5 mg/acetaminophen 325 mg tablet (GRT7014 - Abuse Deterrent Tablet) under fasted conditions.
  Participant must fast from approximately 10:00 pm pre-dosing day until 4 hours after the administration of the Investigational medicinal product (IMP).
  Interventions: Drug: GRT7014 - Abuse Deterrent Tablet
- GRT7014 fed (Experimental): Abuse deterrent formulation of a fixed dose combination of hydrocodone bitartrate 5 mg/acetaminophen 325 mg tablet (GRT7014 - Abuse Deterrent Tablet) under fed conditions.
  Participant must fast from approximately 10:00 pm pre-dosing day until they consume a high-calorie and high-fat breakfast the following morning.
  The IMP must be administered as soon as the meal has been eaten.
  Interventions: Drug: GRT7014 - Abuse Deterrent Tablet
- Norco fasted (Active Comparator): Norco fixed dose combination Hydrocodone bitartrate 5 mg/acetaminophen 325 mg tablet (Norco 5Mg-325Mg Tablet) under fasted conditions.
  Participant must fast from approximately 10:00 pm pre-dosing day until 4 hours after the administration of the IMP.
  Interventions: Drug: Norco 5Mg-325Mg Tablet
- Norco fed (Active Comparator): Norco fixed dose combination Hydrocodone bitartrate 5 mg/acetaminophen 325 mg tablet (Norco 5Mg-325Mg Tablet) under fed conditions.
  Participant must fast from approximately 10:00 pm pre-dosing day until they consume a high-calorie and high-fat breakfast the following morning.
  The IMP must be administered as soon as the meal has been eaten.
  Interventions: Drug: Norco 5Mg-325Mg Tablet

INTERVENTIONS:
Drug: Norco 5Mg-325Mg Tablet — Single oral dose in one of the four cross-over trial periods.
  Other Names: Hydrocodone bitartrate and acetaminophen
  Arms: Norco fasted; Norco fed
Drug: GRT7014 - Abuse Deterrent Tablet — Single oral dose in one of the four cross-over trial periods.
  Other Names: Hydrocodone bitartrate and acetaminophen
  Arms: GRT7014 fasted; GRT7014 fed

SUMMARY:
This clinical trial is being conducted to compare concentrations of hydrocodone and acetaminophen in the blood after administration of a new and a marketed tablet formulation under fasted and fed conditions in healthy adults.

This is a randomized, single-site, open-label, 4-treatment, 4-period crossover, single oral dose Phase I trial in 32 healthy male and female subjects.

The trial will consist of an Enrollment Visit, 4 treatment periods (each lasting approximately 60 hours) separated by 3 washout periods (each lasting at least 7 days), and a Final Examination.

ELIGIBILITY:
Inclusion Criteria:

* Subjects have given written informed consent to participate.
* Body mass index between 20 kg/m2 and 30 kg/m2 inclusive, with a minimum body weight of 60 kg.
* Subjects must be in good health as determined by the medical history, physical and laboratory examinations and must not show any clinically significant deviations from reference ranges as determined by 12-lead electrocardiogram (ECG), vital signs (blood pressure, pulse rate, respiration rate), body temperature, oxygen saturation, and safety laboratory parameters (hematology, clinical chemistry, clotting, and urinalysis).
* From the first administration of IMP until at least the Final Examination, subjects must agree to use highly effective contraception with a low failure rate defined as <1% per year.

For female subjects of childbearing potential:

* Combined (estrogen and progestogen containing) hormonal contraception.
* Progestogen-only hormonal contraception associated with inhibition of ovulation.
* An intra-uterine device (hormone-free).
* An intra-uterine hormone releasing system (IUS).
* Bilateral tubal occlusion.

Women of non-childbearing potential may be included if surgically sterile (i.e., after hysterectomy or bilateral oophorectomy) or post-menopausal for at least 12 months (i.e., spontaneous amenorrhea at least 1 year prior to screening with confirmed follicle-stimulating hormone level >40 IU/L).

For male subjects:

Male subjects have to use barrier contraception (condom) during sexual intercourse with women of childbearing potential from the first application of IMP until the Final Examination. The male subject has to be willing to ensure that the female sexual partner uses at least 1 additional method of contraception with a low failure rate defined as <1% per year.

Exclusion Criteria:

* Withdrawal of informed consent.
* Received forbidden medication or an investigational medical device since the Enrollment Visit.
* Any relevant deterioration in the health of the subject since the Enrollment Visit possibly impacting participation in the trial at the discretion of the investigator, including: adverse events; vital signs (relevant out-of-reference blood pressure or pulse rate if technical failure can be excluded and result is confirmed by at least 1 additional measurement); physical examination, 12-lead ECG (relevant QTc prolongation if result is confirmed by 1 additional ECG measurement and manual re-evaluation by the investigator); other safety parameters.
* Blood loss of 100 mL or more since enrollment in this trial (excluding blood taken for this trial).
* Resting pulse rate <50 beats per minute or >90 beats per minute.
* Resting systolic blood pressure <90 mmHg or >140 mmHg. Resting diastolic blood pressure >90 mmHg.
* Prolongation of corrected QT interval (according to Fridericia's formula; QTcF), i.e., QTcF >450 ms or presence of other of risk factors for torsade de pointes (e.g., heart failure, hypokalemia).
* Evidence for thyroid disease based on clinical and safety laboratory findings, including thyroid stimulating hormone.
* Any laboratory value (from blood samples taken at the Enrollment Visit) meeting the following criteria:

  * Out-of-reference range value for alanine transaminase, aspartate transaminase, alkaline phosphatase, total bilirubin, glucose (fasted), gamma-glutamyl transferase, serum creatinine, prothrombin time, or international normalized ratio.
  * Exclusion range met for urinalysis or lactate dehydrogenase, potassium, total protein, sodium, calcium, hemoglobin, hematocrit, white blood cell count, or platelets.
  * Out-of-reference range value for any other safety laboratory parameter that is judged as clinically relevant by the investigator.
  * A single repeat laboratory test (for each out-of-range parameter) is allowed to rule out laboratory error.
* Positive or missing virus serology test (in blood sample taken at the Enrollment Visit) for human immunodeficiency virus Type 1 or Type 2 antibodies, hepatitis B surface antigen, or hepatitis C virus antibodies.
* For women of childbearing potential only: positive or missing pregnancy test
* Subject received IMP in another clinical trial within 30 days before the Enrollment Visit. Depending on the nature of the previous IMP, a longer washout may be needed.
* Diseases or conditions known to interfere with the absorption, distribution, metabolism, or excretion of drugs.
* History of orthostatic hypotension.
* History of, or at risk of seizures (i.e., head trauma, epilepsy in family history, unclear loss of consciousness).
* Definite or suspected hypersensitivity to the active substance or to any of the excipients of the IMP; especially known hypersensitivity/intolerance or contraindications to opioids (e.g., hydrocodone, hydromorphone), opioid antagonists (e.g., naloxone), acetaminophen or any excipients of the drug formulation.
* Evidence or history of alcohol or drug abuse including positive or missing alcohol breath test or drugs of abuse test.
* Unable to abstain from regular use of any medication, including herbal remedies or over-the-counter medication within 2 weeks prior to the Enrollment Visit and anticipated use during the course of the trial, excluding oral contraceptives in women of childbearing potential and topical medications or nasal sprays without systemic effect.
* Lactating or breastfeeding women.
* Habitually smoking more than 10 cigarettes, 2 cigars, or 2 pipes of tobacco per day within the last 6 months before enrollment in this trial.
* Unable to refrain from smoking for 2 hours before and up to 48 hours after IMP administration in each treatment period, or unable to refrain from smoking as specified in exclusion criterion 16 between 48 hours after IMP and 2 hours before IMP administration in next period.
* Not willing or able to abstain from consumption of:

  * Beverages or food containing methylxanthines (tea, coffee, cola, chocolate, etc.) from 48 hours prior to the planned first administration of IMP until discharge from the trial site in the last treatment period.
  * Beverages or food containing quinine (bitter lemon, tonic water), grapefruit juice (sweet or sour), Seville oranges, or alcohol from 72 hours prior to the planned first administration of IMP until discharge from the trial site in the last treatment period.
* Unwilling or unable to consume a standard high-calorie and high-fat breakfast.
* Known or suspected of not being able to comply with the requirements of the trial protocol or the instructions of the trial site staff.
* Not able to communicate meaningfully with the trial site staff.
* Employee of the investigator or trial site, with direct involvement in the proposed trial or other trials under the direction of that investigator or trial site, as well as family members of the employees or the investigator.
* Blood loss of 500 mL or more (e.g., owing to blood donation) within 45 days before enrollment in this trial.
* Unable to establish reliable venous access.

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 0 (Actual)
Dates: Start 2017-09 (Estimated); Primary Completion 2017-11 (Estimated); Study Completion 2017-11 (Estimated)

PRIMARY OUTCOMES:
Maximum Plasma Concentration (Cmax) | Between 0 hours and 36 hours
  The maximum plasma concentration of hydrocodone and of acetaminophen under fed and fasted conditions.
Area under the plasma concentration curve from timepoint 0 to t (AUC0-t) | Between 0 hours and 36 hours
  The area under the plasma concentration curve of hydrocodone and of acetaminophen under fed and fasted conditions.
Area under the plasma concentration curve from timepoint 0 to infinity (AUC) | Between 0 hours and 36 hours
  The area under the plasma concentration curve of hydrocodone and of acetaminophen under fed and fasted conditions.

CONTACTS AND LOCATIONS:
Overall Officials: Grünenthal Study Director, Study Director — Grünenthal GmbH
Locations (1):
- US001: PRA Health Sciences, Lenexa, Kansas, United States

IPD SHARING:
Plan to Share IPD: No
Details available at:
  http://www.grunenthal.com/grt-web/Grunenthal_Group/Research_Development/Grunenthal_Clinical_Trials/Data_Sharing/296200025.jsp